CLINICAL TRIAL: NCT05361226
Title: The Accuracy of Static Computer-aided Implant Surgery Compared With Conventional Laboratory-guided Implant Surgery for Single-tooth Replacement: A Randomized Controlled Trial
Brief Title: The Accuracy of s-CAIS Compared With c-LIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/DT071-1
Record Dates: First submitted 2022-04-10; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Dental Implant
Keywords: Clinical Research; static computer aided implant surgery; accuracy; Dental implant
MeSH Terms: interventions — Dimensional Measurement Accuracy

STUDY DESIGN:
Intervention Model Description: Forty participants were allocated to two study groups via the coin-tossing technique.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- s-CAIS (static computer aided implant surgery) (Experimental): For the s-CAIS group, Cone Beam Computed Tomography (CBCT) and full-arch optical scan were performed to provide digital information for implant planning software (coDiagnostix 9, Dental Wings GmbH, Chemnitz, Germany). The virtual implant was set on a three dimensional (3D) virtual jaws according to the prosthetically driven protocol by one postgraduate dentist and was confirmed by one experienced dentist. Static surgical template covering on occlusal part of 4 teeth anteroposteriorly was then fabricated via 3D printing machine (surgical guide resin, Form 2, Formlabs, Somerville, Massachusetts, USA). This surgical template would be used during surgery.
  Interventions: Other: Accuracy measurement
- c-LIS (conventional laboratory-guided implant surgery) (Active Comparator): For the c-LIS group, a radiographic template (ORTHO Plast, prominent®, Chonburi, Thailand) was fabricated covering on occlusal part of 4 teeth anteroposteriorly according to diagnostic wax-up on the study model. A radiographic marker (gutta percha) was then filled in the created hole of the template and for used while taking CBCT image to verify marker position.
  Next, a study model was scanned by laboratory surface scan (D900m, 3Shape, Copenhagen, Denmark). The STL file was imported to 3D printing devices and the resin model was fabricated (Dental LT clear resin, Form 2, Formlabs, Somerville, Massachusetts, USA).
  Next, the same template that had been used for CBCT was used to place implant replicas in a resin model. The position of the implant replicas in the models were assumed as pre-operative planned implant position.
  Interventions: Other: Accuracy measurement

INTERVENTIONS:
Other: Accuracy measurement — Three months following the implant placement, patients were called back to the implant clinic to record the actual implant position with the digital impression technique. Full mouth scans were done by using the intraoral scanner (Trios 3, 3Shape, Copenhagen, Denmark). The surface scans were then exported as an STL file and were imported to coDiagnostiX software. The "Treatment evaluation tool" function tool was used to measure the accuracy of the implant placement which measured the amount of deviation of the placed implant from the planned position. The outcomes were generated into three main parameters.

SUMMARY:
To compare the static computer-aided implant surgery (s-CAIS) and conventional laboratory-guided implant surgery (c-LIS) in terms of accuracy for single tooth replacement in posterior areas.

DETAILED DESCRIPTION:
There was still a lack of evidence in randomized clinical studies about the accuracy measurement comparing digital and laboratory workflows with tooth-supported templates for single implant cases in the posterior regions. Therefore, this present study's primary investigation was to perform accuracy measurement comparing digital and laboratory workflows with tooth-supported templates for single implant cases in the posterior regions. The secondary investigation was to find the effect of several factors on the accuracy of implant placement in these areas.

ELIGIBILITY:
Inclusion Criteria:

* Patients had a partially edentulous ridge in the premolar-molar region with existing two-sided interproximal as well as antagonistic contacts
* Patients had healthy periodontal status and adequate keratinized gingiva at the edentulous space

Exclusion Criteria:

* - Patients have any local and systemic diseases considered as contraindications for dental implant treatment.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The accuracy of implant placement | Three months after implant placement
  Patients were called back to record the actual implant position with the the intraoral scanner (Trios 3, 3Shape, Copenhagen, Denmark). The surface scans were then exported as an STL file and were imported to coDiagnostiX software. Those postoperative surface scans were merged with the preoperative surface scan in each group protocols. The "Treatment evaluation tool" function tool was used to measure the accuracy of the implant placement which measured the amount of deviation of the placed implant from the planned position. The outcomes were generated into three main parameters which were Angular deviation, Coronal global deviation and Apical global deviation.
  Angular deviation = the amount of angle(°), in which the actually placed implant deviated from the virtually planned implant in 3D.
  Coronal/ Apical global deviation = the amount of distance(mm), in which the actually placed implant deviated from the virtually planned implant at the coronal/ apical position in 3D.

SECONDARY OUTCOMES:
Factors influencing the accuracy of implant placement | Three months after implant placement
  Various factors influencing the accuracy of implant placement were also analyzed including the type of arch (Maxilla vs. Mandible), side of the arch (Left vs. Right), implant location (Premolar vs. Molar), implant diameter (WN vs. RN), implant length (8 vs. 10 mm), ridge morphology (Broad (≥8mm) vs. Narrow (˂8mm), cortical bone thickness and cortical interference. The thickness of the cortical bone was evaluated at the center of the implant after the planned implant position was completely set in the coDiagnostiX program. If any parts of the planned implant involving against any cortical bone walls, it would count as having a cortical interference.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jung RE, Schneider D, Ganeles J, Wismeijer D, Zwahlen M, Hammerle CH, Tahmaseb A. Computer technology applications in surgical implant dentistry: a systematic review. Int J Oral Maxillofac Implants. 2009;24 Suppl:92-109. PMID 19885437
- [Background] D'haese J, Ackhurst J, Wismeijer D, De Bruyn H, Tahmaseb A. Current state of the art of computer-guided implant surgery. Periodontol 2000. 2017 Feb;73(1):121-133. doi: 10.1111/prd.12175. PMID 28000275
- [Background] Hultin M, Svensson KG, Trulsson M. Clinical advantages of computer-guided implant placement: a systematic review. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:124-35. doi: 10.1111/j.1600-0501.2012.02545.x. PMID 23062137
- [Background] Younes F, Eghbali A, De Bruyckere T, Cleymaet R, Cosyn J. A randomized controlled trial on the efficiency of free-handed, pilot-drill guided and fully guided implant surgery in partially edentulous patients. Clin Oral Implants Res. 2019 Feb;30(2):131-138. doi: 10.1111/clr.13399. Epub 2019 Jan 7. PMID 30578650
- [Background] Behneke A, Burwinkel M, Behneke N. Factors influencing transfer accuracy of cone beam CT-derived template-based implant placement. Clin Oral Implants Res. 2012 Apr;23(4):416-23. doi: 10.1111/j.1600-0501.2011.02337.x. Epub 2011 Oct 24. PMID 22092586
- [Background] Cassetta M, Stefanelli LV, Giansanti M, Calasso S. Accuracy of implant placement with a stereolithographic surgical template. Int J Oral Maxillofac Implants. 2012 May-Jun;27(3):655-63. PMID 22616060
- [Background] Zhao XZ, Xu WH, Tang ZH, Wu MJ, Zhu J, Chen S. Accuracy of computer-guided implant surgery by a CAD/CAM and laser scanning technique. Chin J Dent Res. 2014;17(1):31-6. PMID 25028687
- [Background] Tahmaseb A, Wu V, Wismeijer D, Coucke W, Evans C. The accuracy of static computer-aided implant surgery: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:416-435. doi: 10.1111/clr.13346. PMID 30328191
- [Background] Gallardo YNR, da Silva-Olivio IR, Gonzaga L, Sesma N, Martin W. A Systematic Review of Clinical Outcomes on Patients Rehabilitated with Complete-Arch Fixed Implant-Supported Prostheses According to the Time of Loading. J Prosthodont. 2019 Dec;28(9):958-968. doi: 10.1111/jopr.13104. Epub 2019 Oct 18. PMID 31433096
- [Background] Geng W, Liu C, Su Y, Li J, Zhou Y. Accuracy of different types of computer-aided design/computer-aided manufacturing surgical guides for dental implant placement. Int J Clin Exp Med. 2015 Jun 15;8(6):8442-9. eCollection 2015. PMID 26309497
- [Background] Pozzi A, Polizzi G, Moy PK. Guided surgery with tooth-supported templates for single missing teeth: A critical review. Eur J Oral Implantol. 2016;9 Suppl 1:S135-53. PMID 27314119
- [Background] Tahmaseb A, Wismeijer D, Coucke W, Derksen W. Computer technology applications in surgical implant dentistry: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:25-42. doi: 10.11607/jomi.2014suppl.g1.2. PMID 24660188
- [Background] Di Giacomo GA, Cury PR, de Araujo NS, Sendyk WR, Sendyk CL. Clinical application of stereolithographic surgical guides for implant placement: preliminary results. J Periodontol. 2005 Apr;76(4):503-7. doi: 10.1902/jop.2005.76.4.503. PMID 15857088
- [Background] Ersoy AE, Turkyilmaz I, Ozan O, McGlumphy EA. Reliability of implant placement with stereolithographic surgical guides generated from computed tomography: clinical data from 94 implants. J Periodontol. 2008 Aug;79(8):1339-45. doi: 10.1902/jop.2008.080059. PMID 18672982
- [Background] Choi W, Nguyen BC, Doan A, Girod S, Gaudilliere B, Gaudilliere D. Freehand Versus Guided Surgery: Factors Influencing Accuracy of Dental Implant Placement. Implant Dent. 2017 Aug;26(4):500-509. doi: 10.1097/ID.0000000000000620. PMID 28731896
- [Background] Farley NE, Kennedy K, McGlumphy EA, Clelland NL. Split-mouth comparison of the accuracy of computer-generated and conventional surgical guides. Int J Oral Maxillofac Implants. 2013 Mar-Apr;28(2):563-72. doi: 10.11607/jomi.3025. PMID 23527361
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509
- [Background] Kunavisarut C, Santivitoonvong A, Chaikantha S, Pornprasertsuk-Damrongsri S, Joda T. Patient-reported outcome measures comparing static computer-aided implant surgery and conventional implant surgery for single-tooth replacement: A randomized controlled trial. Clin Oral Implants Res. 2022 Mar;33(3):278-290. doi: 10.1111/clr.13886. Epub 2022 Jan 2. PMID 34921690
- [Background] Buser D, Martin W, Belser UC. Optimizing esthetics for implant restorations in the anterior maxilla: anatomic and surgical considerations. Int J Oral Maxillofac Implants. 2004;19 Suppl:43-61. PMID 15635945
- [Background] Buser D, Chappuis V, Kuchler U, Bornstein MM, Wittneben JG, Buser R, Cavusoglu Y, Belser UC. Long-term stability of early implant placement with contour augmentation. J Dent Res. 2013 Dec;92(12 Suppl):176S-82S. doi: 10.1177/0022034513504949. Epub 2013 Oct 24. PMID 24158332
- [Background] Tarnow DP, Cho SC, Wallace SS. The effect of inter-implant distance on the height of inter-implant bone crest. J Periodontol. 2000 Apr;71(4):546-9. doi: 10.1902/jop.2000.71.4.546. PMID 10807116
- [Background] Tolstunov L. Classification of the alveolar ridge width: implant-driven treatment considerations for the horizontally deficient alveolar ridges. J Oral Implantol. 2014 Jul;40 Spec No:365-70. doi: 10.1563/aaid-joi-D-14-00023. Epub 2014 Feb 27. PMID 24575743
- [Background] Derksen W, Wismeijer D, Flugge T, Hassan B, Tahmaseb A. The accuracy of computer-guided implant surgery with tooth-supported, digitally designed drill guides based on CBCT and intraoral scanning. A prospective cohort study. Clin Oral Implants Res. 2019 Oct;30(10):1005-1015. doi: 10.1111/clr.13514. Epub 2019 Sep 9. PMID 31330566
- [Background] Nokar S, Moslehifard E, Bahman T, Bayanzadeh M, Nasirpouri F, Nokar A. Accuracy of implant placement using a CAD/CAM surgical guide: an in vitro study. Int J Oral Maxillofac Implants. 2011 May-Jun;26(3):520-6. PMID 21691598
- [Background] Sarment DP, Sukovic P, Clinthorne N. Accuracy of implant placement with a stereolithographic surgical guide. Int J Oral Maxillofac Implants. 2003 Jul-Aug;18(4):571-7. PMID 12939011
- [Background] Smitkarn P, Subbalekha K, Mattheos N, Pimkhaokham A. The accuracy of single-tooth implants placed using fully digital-guided surgery and freehand implant surgery. J Clin Periodontol. 2019 Sep;46(9):949-957. doi: 10.1111/jcpe.13160. Epub 2019 Jul 19. PMID 31241782
- [Background] Park JY, Song YW, Park SH, Kim JH, Park JM, Lee JS. Clinical factors influencing implant positioning by guided surgery using a nonmetal sleeve template in the partially edentulous ridge: Multiple regression analysis of a prospective cohort. Clin Oral Implants Res. 2020 Dec;31(12):1187-1198. doi: 10.1111/clr.13664. Epub 2020 Sep 22. PMID 32905643
- [Background] Cassetta M, Di Mambro A, Giansanti M, Stefanelli LV, Cavallini C. The intrinsic error of a stereolithographic surgical template in implant guided surgery. Int J Oral Maxillofac Surg. 2013 Feb;42(2):264-75. doi: 10.1016/j.ijom.2012.06.010. Epub 2012 Jul 11. PMID 22789635
- [Background] Schneider D, Marquardt P, Zwahlen M, Jung RE. A systematic review on the accuracy and the clinical outcome of computer-guided template-based implant dentistry. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:73-86. doi: 10.1111/j.1600-0501.2009.01788.x. PMID 19663953
- [Background] El Kholy K, Lazarin R, Janner SFM, Faerber K, Buser R, Buser D. Influence of surgical guide support and implant site location on accuracy of static Computer-Assisted Implant Surgery. Clin Oral Implants Res. 2019 Nov;30(11):1067-1075. doi: 10.1111/clr.13520. Epub 2019 Aug 20. PMID 31381178
- [Background] El Kholy K, Janner SFM, Schimmel M, Buser D. The influence of guided sleeve height, drilling distance, and drilling key length on the accuracy of static Computer-Assisted Implant Surgery. Clin Implant Dent Relat Res. 2019 Feb;21(1):101-107. doi: 10.1111/cid.12705. Epub 2018 Dec 27. PMID 30589502
- [Background] Pettersson A, Kero T, Gillot L, Cannas B, Faldt J, Soderberg R, Nasstrom K. Accuracy of CAD/CAM-guided surgical template implant surgery on human cadavers: Part I. J Prosthet Dent. 2010 Jun;103(6):334-42. doi: 10.1016/S0022-3913(10)60072-8. PMID 20493322
- [Background] Vieira DM, Sotto-Maior BS, Barros CA, Reis ES, Francischone CE. Clinical accuracy of flapless computer-guided surgery for implant placement in edentulous arches. Int J Oral Maxillofac Implants. 2013 Sep-Oct;28(5):1347-51. doi: 10.11607/jomi.3156. PMID 24066327
- [Background] Van Assche N, Vercruyssen M, Coucke W, Teughels W, Jacobs R, Quirynen M. Accuracy of computer-aided implant placement. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:112-23. doi: 10.1111/j.1600-0501.2012.02552.x. PMID 23062136
- [Background] Ozan O, Orhan K, Turkyilmaz I. Correlation between bone density and angular deviation of implants placed using CT-generated surgical guides. J Craniofac Surg. 2011 Sep;22(5):1755-61. doi: 10.1097/SCS.0b013e31822e6305. PMID 21959426
- [Background] Cushen SE, Turkyilmaz I. Impact of operator experience on the accuracy of implant placement with stereolithographic surgical templates: an in vitro study. J Prosthet Dent. 2013 Apr;109(4):248-54. doi: 10.1016/S0022-3913(13)60053-0. PMID 23566606
- [Background] Rungcharassaeng K, Caruso JM, Kan JY, Schutyser F, Boumans T. Accuracy of computer-guided surgery: A comparison of operator experience. J Prosthet Dent. 2015 Sep;114(3):407-13. doi: 10.1016/j.prosdent.2015.04.004. Epub 2015 Jun 25. PMID 26119019
- [Background] Sugiura T, Yamamoto K, Horita S, Murakami K, Tsutsumi S, Kirita T. The effects of bone density and crestal cortical bone thickness on micromotion and peri-implant bone strain distribution in an immediately loaded implant: a nonlinear finite element analysis. J Periodontal Implant Sci. 2016 Jun;46(3):152-65. doi: 10.5051/jpis.2016.46.3.152. Epub 2016 Jun 28. PMID 27382504